CLINICAL TRIAL: NCT01328392
Title: Evaluating Treatment Response in Laryngo-Pharyngeal Reflux
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The sponsor did not fund the study.
Sponsor: University of Washington (Other)
Collaborators: Takeda Pharmaceuticals North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 39853
Record Dates: First submitted 2011-03-30; First posted 2011-04-04 (Estimated); Last update posted 2017-07-05 (Actual); Status verified 2011-03

CONDITIONS: Laryngo-pharyngeal Reflux
Keywords: LPR; GERD
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Dexlansoprazole

INTERVENTIONS:
Drug: Dexlansoprazole — 30mg a day, 3 months
  Other Names: Dexilant

SUMMARY:
Although laryno-pharyngeal reflux (LPR) and gastroesophageal reflux disease (GERD) differ in symptoms and treatment, they are diagnosed by the same standard 24-hour pH monitoring system which measures liquid reflux in the esophagus. The investigators are evaluating a new 24-hour pharyngeal pH monitoring system by Restech which can measure acid exposure in the airway and can be used specifically for LPR diagnosis. The purpose of this study is to determine whether the Restech device is more effective than standard pH monitoring in predicting the response to proton pump inhibitor (PPI) acid suppression therapy using Dexlansoprazole in patients with symptoms and/or manifestations of LPR.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years old or above
* Have a clinical diagnosis of LPR
* Able and willing to provide consent

Exclusion Criteria:

* History of any previous anti-reflux operation or procedure
* History of pharyngeal or laryngeal surgery
* History of larngeal or hypolaryngeal neoplasm
* Allergy or significant adverse reaction to PPI
* Patient on PPI therapy within 4 weeks prior to enrollment
* A cumulative history of PPI therapy equal to or greater than 3 months
* History of noncompliance with medication or study protocols
* Enrolled in another clinical trial using investigational medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-05; Primary Completion 2012-04 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Ability of Restech to predict LPR symptom improvement after treatment with Dexlansoprazole. | 3 months
  Successful LPR symptom improvement will be defined as a 25% improvement in Reflux Symptom Index (RSI)after 3 months of Dexlansoprazole.

SECONDARY OUTCOMES:
Comparison between standard pH data and Restech data (normal vs.abnormal acid exposure, using established normative data values) before and after treatment with Dexlansoprazole. | 3 months
Correlation between Restech acid exposure events and standard pH monitoring acid exposure events. | 3 months
  Using a method similar to the calculation of a symptom index for each study in each patient, to determine the percentage of time in which a Restech-detected acid event occurs at the same time as an acid event detected on standard pH monitoring.
Laryngoscopic findings pre and post Dexlansoprazole treatment. | 3 months
  Expressed as Reflux Finding Score (RFS).
Differences between RSI and general GERD symptom questionnaire scores on and off Dexlansoprazole. | 3 months
Correlation of RSI and general GERD symptom questionnaire scores with Restecha dn standard pH values. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Brant K Oelschlager, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States